CLINICAL TRIAL: NCT03111277
Title: Phase 1 Clinical Trial for MR Guided Focused Ultrasound (FUS) Thalamotomy of Central Lateral Thalamic Nucleus for the Treatment of Neuropathic Pain
Brief Title: MR Guided Focused Ultrasound for Treatment of Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Focused Ultrasound Foundation (Other); InSightec (Industry)
Responsible Party: Principal Investigator, Dheeraj Gandhi, Professor of Radiology, Neurology and Neurosurgery, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HP-00068223
Record Dates: First submitted 2017-03-27; First posted 2017-04-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Severe Neuropathic Pain Due to Radiculopathy or Radicular Injury; Spinal Cord Injuries; Phantom Limb Pain
Keywords: neuropathic pain
MeSH Terms: conditions — Spinal Cord Injuries; Phantom Limb; Neuralgia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental: ExAblate Transcranial treatment (Experimental): The ExAblate Transcranial system will be used to destroy a small cluster of cells that may be causing the study participant's pain . The ExAblate uses ultrasound to heat a small spot in the brain. Ultrasound passes through the skin and skull and into the brain to focus on a spot the study investigator wants to treat.
  Interventions: Device: Experimental: ExAblate Transcranial treatment

INTERVENTIONS:
Device: Experimental: ExAblate Transcranial treatment — Patients' head will be placed in a device to hold it still for the treatment. Patients will lie headfirst on the ExAblate table. The ExAblate Transcranial helmet will be placed on their head. A device will be placed over their head to hold it and the helmet still. The investigators will measure the study participant's heart, blood pressure, temperature, and breathing rate before the treatment begins. MRI scans will be taken to make sure the ultrasound waves will be aimed exactly within the target. The space between the rubber diaphragm and the helmet will be filled with water. The water will be chilled to avoid heating of the scalp and skull during the ultrasound treatment. A series of MR images will be taken to identify the target area, and plan the study treatment. The study investigators will decide on the area of participant's brain that will be treated. The ExAblate Transcranial system will compute a plan to cover the treatment area.
  Other Names: The ExAblate® MR guided focused ultrasound system

SUMMARY:
Neuropathic pain is often a result of direct diseases of peripheral or central nervous system with an estimated prevalence of 8% of adults and this pain is associated with significant consequences because of longer symptom duration and severity than many of the other pain syndromes. Functional brain imaging has revealed that many regions of the brain are engaged by painful events, but specific areas such as the thalamus have been markedly implicated.

The purpose of this study is to determine the feasibility and safety of MRI-guided focused ultrasound treatment using the ExAblate Transcranial System in patients suffering from Neuropathic pain. This treatment modality offers non-invasive precise treatment potential for these patients.

DETAILED DESCRIPTION:
The primary purpose of this study is to assess the safety of MRI-guided focused ultrasound (MRgFUS) in patients with chronic neuropathic pain whose medicines are not working well. The device that will be used to create and send ultrasound waves through the skull is called the ExAblate Transcranial system. The ultrasounds waves will precisely target a small part of the brain known as the thalamus. Chronic neuropathic pain is a common type of disabling pain that affects people.

Usually, people with chronic neuropathic pain are treated with medicines to control the pain. However, these medications may not provide adequate relief of the pain or may be associated with undesirable side effects. This study intends to investigate the use of a new technology The ExAblate transcranial system for treating patients that are not responding to medications and continue to have disabling pain.

The ExAblate Transcranial system will be used to destroy a small cluster of cells that may be causing the study participant's pain . The ExAblate uses ultrasound to heat a small spot in the brain. The process of ablation is similar to a magnifying glass that uses light to heat a small spot on a piece of paper. Ultrasound passes through the skin and skull and into the brain to focus on a spot the study investigator wants to treat.Once the spot is destroyed, it cannot grow back.

ELIGIBILITY:
Inclusion Criteria:

* These include patients with:

  1. Severe uncontrolled neuropathic pain due to radiculopathy or radicular injury
  2. Spinal Cord Injury
  3. Phantom Limb Pain

Patients that have had prior motor cortex stimulation or spinal cord stimulators will be eligible provided that the hardware has been removed at least six months ago. Detailed inclusion and exclusion criteria for the study are listed below:

Inclusion criteria:

1. Age greater than 21 and less than 75 years
2. Subjects who are able and willing to give consent and able to attend all study visits,
3. Documented Neuropathic pain for more than 6 months duration, confirmed from clinical history and examination by a pain specialist or neurologist
4. Failure to respond to any of the usual therapeutic regimens considered to be standard of care for neuropathic pain. The patient should have failed a trial of at least three pain medications, including at least one opioid agent
5. Patients with radiculopathy or radicular injury or phantom limb pain should have failed one additional pain intervention such as nerve block, epidural steroid injection, motor cortex or spinal cord stimulator
6. Patients with Spinal cord injury, in addition to having failed a trial of three pain medications, should have failed one additional intervention such as Botox injection or intra-thecal baclofen.
7. Subjects should have been on stable dose of analgesic agents for at least a period of 4 weeks
8. Clinical symptoms consistent with persistent, intractable pain that has remained at average NRS score >5 for 30 days, significant pain related disability (Pain Disability Index (PDI) score >30) or severe allodynia.
9. Central lateral thalamotomy is feasible based on evaluation of imaging studies
10. Patient able to communicate sensations during the ExAblate TcMRgFUS treatment
11. Two members of the medical team have agreed upon inclusion and exclusion criteria.

Exclusion Criteria:

1. Patient with contra-indications to MRI such as severe claustrophobia and metallic implants incompatible with MRI.
2. Severe psychiatric disorder such as uncontrolled depression, bipolar disorder, prior attempt at suicide or suicide ideation in preceding 12 months
3. Life expectancy less than 12 months
4. Anticoagulant or antiplatelet medications as well as underlying coagulopathy
5. Prior or currently implanted thalamic DBS
6. Pregnant ladies or women of childbearing age who are sexually active and not using contraception
7. Inability to provide informed consent, for example due to underlying cognitive impairment or aphasia
8. Presence of intracranial mass or an acute intracranial abnormality
9. Subjects with unstable cardiac status such as Unstable angina pectoris, documented myocardial infarction within 6 months of protocol entry and ejection fraction less than 40
10. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within a 12 month period:

    1. Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household).
    2. Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
    3. Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
    4. Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights).
11. Severe hypertension (diastolic BP > 100 on medication or persistently elevated SBP>140 mmHg despite antihypertensive medications)
12. History of immunocompromise including those who are HIV positive.
13. History of CNS disease (this includes but not limited to intracranial hemorrhage, Traumatic brain injury or thalamic stroke, seizures within the past year, brain tumors, multiple CVA or CVA within 6 months)
14. Subjects with life-threatening systemic disease that include and not limited to the following will be excluded from the study participation: HIV, Liver Failure, blood dyscrasias, etc.
15. Individuals who are not able or willing to tolerate the required prolonged stationary supine position during treatment (can be up to 4 hrs of total table time.)
16. Are participating or have participated in another clinical trial in the last 30 days
17. Patients receiving a Morphine equivalent dose of greater than 90 mg per day
18. Subjects who have non-neuropathic pain as the major component of their pain presentation will be excluded from the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2022-10-09 (Actual); Study Completion 2022-10-09 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment related adverse events | All events will be reported upto 12 months from treatment
  Procedure related or device related adverse events will be reported, from the treatment day through the 12-month follow-up period.

SECONDARY OUTCOMES:
Change in pain measurements using pain numeric rating scale | 12 months
  Reduction at 12 months in maximum or average pain scores as measured on Pain numeric rating scale (NRS) by 40% or more without increase in medication consumption by more than 25%.
Change in pain related disability | 12 months
  Reduction in Pain related disability by greater than or equal to 30% using pain interference scale on the Brief pain inventory (BPI) at 12-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dheeraj Gandhi, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland School of Medicine and University of Maryland Medical Systems, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Ahmed AK, Zhuo J, Gullapalli RP, Jiang L, Keaser ML, Greenspan JD, Chen C, Miller TR, Melhem ER, Sansur CA, Eisenberg HM, Gandhi D. Focused Ultrasound Central Lateral Thalamotomy for the Treatment of Refractory Neuropathic Pain: Phase I Trial. Neurosurgery. 2024 Apr 1;94(4):690-699. doi: 10.1227/neu.0000000000002752. Epub 2023 Nov 10. PMID 37947407